CLINICAL TRIAL: NCT01193114
Title: Stage 1 Treatment Development With Homeless Mothers and Their 2-6 Year Old Children
Brief Title: Stage 1 Treatment Development With Homeless Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Natasha Slesnick, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008B0309; R01DA023908 (NIH)
Record Dates: First submitted 2010-02-02; First posted 2010-09-01 (Estimated); Results first posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-01

CONDITIONS: Substance Abuse
Keywords: substance abuse; homeless mothers
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ecologically-Based Behavioral Treatment (Experimental): Ecologically-Based Treatment was provided over a period of 6 months. The treatment integrated independent housing, case management services and substance abuse counseling. Specifically, the mothers were housed in an apartment of their choice and received three months of utility and rental assistance of up to $600 per month.
  Interventions: Behavioral: Ecologically Based Treatment (EBT)
- Treatment as Usual (Active Comparator): The Mothers were offered services provided through the family shelter.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Ecologically Based Treatment (EBT) — Substance abuse treatment (the Community Reinforcement Approach), case management and housing.
  Arms: Ecologically-Based Behavioral Treatment
Behavioral: Treatment as Usual (TAU) — Treatment/intervention as normally provided by community service agencies that service substance abusing homeless families.
  Arms: Treatment as Usual

SUMMARY:
Aim 1. Identify specific targets and processes of intervention among homeless substance abusing mothers with children between the ages of 2 and 6 years from information collected in focus groups and assessment interviews. Translate that information for the refinement of the ecologically based treatment manual.

Aim 2. Test the efficacy of the treatment in a nonrandomized pilot study and revise the manual based upon those findings.

Aim 3. Test the efficacy of the experimental intervention compared to treatment as usual (TAU) in a randomized pilot, with the goal to improve maternal substance abuse problems, social stability, and mental health. It is expected that the experimental intervention will be associated with lower substance use and related problem behaviors than TAU.

Aim 4. Test whether intended change processes (mediators) associated with the intervention produce the desired change in mother's substance use, social stability, and mental health. It is expected that self-efficacy will mediate substance use outcomes.

Aim 5. Explore how length of homelessness, age and ethnicity of the mother predict treatment response (moderators).

Aim 6. Explore the impact of the experimental intervention (Ecologically-Based Therapy)on interpersonal stress and child's mental health.

DETAILED DESCRIPTION:
Even with increased focus on those experiencing homelessness, the number of homeless families continues to rise, with the demand for temporary shelter so high that many cities are unable to meet the needs of these families. The majority of these families are headed by single mothers, many of whom struggle with substance use and mental health issues. These struggles are in addition to meeting the basic needs of themselves and their children. No study has documented an effective approach for intervening with homeless substance abusing mothers with children. Research attention towards identifying efficacious interventions for this population which address the multiple needs of these families is thus considered an important focus for reducing significant individual and social costs associated with substance use and homelessness. The current study utilizes an ecological systems approach as the theoretical base for the proposed treatment. The overarching goals of the current treatment development study are to first identify targets and processes of intervention desired by homeless mothers and then pilot test a novel manualized intervention focused on improving treatment success of this special population. In Stage 1a, information from the multi-method assessment and focus groups with N=30 homeless mothers will guide modifications to an integrated intervention that includes housing, case management and the Community Reinforcement Approach. The final manual resulting from this important study will address the multiple needs of homeless mothers, including basic needs and substance use/mental health problems. The intervention will be tested in a nonrandomized pilot (N = 15) in which interview and self-report methods will be used for data gathering. Follow-up will be conducted at 3 and 6 months post baseline and the intervention will be modified based upon the process and outcome analyses. Finally, the revised intervention will be tested in Stage 1b in a randomized pilot study involving 60 women and children assigned to the project intervention (N = 30) or treatment as usual (N=30) and followed at 3, 6, and 9 months post-baseline. In the randomized pilot study an effect size will be computed for use in informing a larger, randomized Stage II trial. This project utilizes existing efficacious models of drug abuse treatment to generate valuable new information critical to treatment services delivery for a special population of substance abusers. Since homeless substance abusing women and their children are at increased risk for a variety of adverse outcomes, improved maternal and child outcomes may produce substantial health-care benefits to the women, their children, and society at large. The findings from this study will serve as the foundation for the refinement and implementation of a promising intervention for drug-addicted homeless women and children that can then be tested for efficacy in a Stage II trial.

ELIGIBILITY:
Inclusion Criteria:

* residing at a homeless shelter for families
* meet diagnostic criteria for psychoactive substance use or alcohol disorder
* has physical custody of a biological child between the ages of 2 to 6 years old

Exclusion Criteria:

* evidence of unremitted psychosis or other condition that would impair the mothers' ability to understand and participate in the intervention research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Slesnick, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Department of Human Development and Family Science, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.60 (5.54) | 27 (6.46) | 26.30 (6.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percent Days of Substance Use in the Prior 3 Months.
Time Frame: 3 months post-baseline measure
Population: The analysis was conducted with all of the collected data. Discrepancies in number of participants between the Participant Flow Module and the analysis are due to missing data.
Measure: Mean (Standard Deviation); unit: percent days of substance use
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual
Number analyzed (Participants) | 30 | 24
percent days of substance use | 45.40 (38.79) | 49.17 (41.87)

2. Primary Outcome: Percent Days of Substance Use in the Prior 3 Months.
Time Frame: 6 months post-baseline measure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent days of substance use
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual
Number analyzed (Participants) | 30 | 23
percent days of substance use | 34.55 (39.09) | 46.84 (36.29)

3. Primary Outcome: Percent Days of Substance Use in the Prior 3 Months.
Time Frame: 9 months post-baseline measure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent days of substance use
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual
Number analyzed (Participants) | 30 | 24
percent days of substance use | 41.74 (38.53) | 44.54 (41.67)

4. Secondary Outcome: BDI Depression Score
Description: Beck Depression Inventory - II (BDI - II) Range from 0 (no depression) to 63 (severe depression)
Time Frame: 3 months post-baseline measure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual
Number analyzed (Participants) | 30 | 24
units on a scale | 15.03 (15.10) | 13.63 (10.03)

5. Secondary Outcome: BDI Depression Score
Description: Beck Depression Inventory - II (BDI - II) Range from 0 (no depression) to 63 (severe depression)
Time Frame: 6 months post-baseline measure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual
Number analyzed (Participants) | 30 | 23
units on a scale | 14.63 (13.67) | 14.91 (11.17)

6. Secondary Outcome: BDI Depression Score
Description: Beck Depression Inventory - II (BDI - II) Range from 0 (no depression) to 63 (severe depression)
Time Frame: 9 months post-baseline measure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual
Number analyzed (Participants) | 29 | 24
units on a scale | 13.21 (13.46) | 13.38 (12.06)

ADVERSE EVENTS:
Time Frame: Overall Study
Description: Adverse events were monitored but none were observed.
Arm/Group | Ecologically-Based Behavioral Treatment | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No